CLINICAL TRIAL: NCT07200752
Title: Effects of Telerehabilitation Versus Supervised Physiotherapy on Neck Muscle Endurance, Pain, and Disability in KARABUK University Students With Text Neck Syndrome: A Randomized Controlled Trial
Brief Title: Effects of Exercise Training Delivered Through Telerehabilitation on Text Neck Syndrome
Acronym: TEXT NECK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, PT, PhD, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBU TEXT NECK
Record Dates: First submitted 2025-09-19; First posted 2025-10-01 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Text Neck Syndrome; Telerehabilitation; Exercise
Keywords: TEXT NECK; PAIN MANEGMENT; NECK MUSCLE ENDURANCE; TELEREHABILITATION
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitaion exercise program (Experimental): telerehabilitation based neck exercise training
  Interventions: Behavioral: Telerehabilitation-Based Neck Exercise Training
- supervised in-person exercise program (Active Comparator): supervised physiotherapy exercise training
  Interventions: Behavioral: Supervised physiotherapy exercise training

INTERVENTIONS:
Behavioral: Telerehabilitation-Based Neck Exercise Training — Participants received a 6-week Telerehabilitation exercise program delivered via video calls and digital platforms, three sessions per week. The program included stretching, active range of motion, isometric strengthening, and postural correction exercises with progressive intensity.
  Arms: Telerehabilitaion exercise program
Behavioral: Supervised physiotherapy exercise training — Participants received the same 6-week exercise program as the Telerehabilitation group, but delivered face-to-face in a supervised clinical setting by a physiotherapist, three sessions per week.
  Arms: supervised in-person exercise program

SUMMARY:
To compare the effectiveness of telerehabilitation exercise program with that of supervised in-person physiotherapy in improving neck muscle endurance, pain intensity, and functional disability in university students with text neck syndrome. Methods:

A randomized controlled trial was conducted with 31 university students aged 18-24 diagnosed with text neck syndrome. Participants were randomly assigned to either a telerehabilitation group or a supervised in-person exercise group. Both groups received an identical six-week exercise program, delivered three times per week, including stretching, range of motion, isometric, and postural correction exercises with progressive intensity. Primary outcomes included deep cervical flexor and extensor muscle endurance. Secondary outcomes were neck pain intensity and functional disability. Assessments were performed at baseline and post-intervention.

DETAILED DESCRIPTION:
Introduction

Text Neck Syndrome, also known as turtle neck posture, is a repetitive stress injury of the neck associated with prolonged use of handheld electronic devices that disrupts cervical spine alignment and function. When users maintain a forward head posture, particularly while using smartphones, this can lead to upper back discomfort, muscle spasms, shoulder stiffness, and cramps due to increased mechanical load on cervical tissues. The term Text Neck was introduced to describe this phenomenon. Biomechanical modeling has shown that as cervical flexion increases, the mechanical load on the cervical spine rises substantially, which can encourage loss of the natural cervical curvature and promote kyphotic changes in the upper thoracic spine. These postural alterations may destabilize ergonomics and contribute to musculoskeletal dysfunction. If left untreated, text neck posture may result in long-term structural changes, including vertebral misalignment, neuromuscular impairment, and chronic pain syndromes. Additionally, abnormal head posture is associated with impaired proprioception, increased postural sway, and reduced balance control. Telerehabilitation, defined as the delivery of therapeutic interventions through digital platforms, offers a promising alternative to in-person therapy by overcoming barriers related to distance, mobility, and cost. Its widespread adoption during the COVID-19 pandemic demonstrated that remotely supervised neck exercise programs can produce results comparable to traditional care for chronic neck pain. Telerehabilitation has been associated with reduced pain intensity, improved physical function, and enhanced quality of life in individuals experiencing neck pain.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

Participants will be eligible for inclusion if they meet all of the following criteria:

Are between 18 and 24 years of age.

Report smartphone use exceeding 3 hours per day.

Present with at least three of the following symptoms:

Neck pain

Shoulder pain

Upper back pain

Headache

Insomnia

Tingling or numbness in the hands

All participants will be screened for eligibility by a licensed physiotherapist, and only those who meet all inclusion and none of the exclusion criteria will be randomized.

Exclusion Criteria:

Participants will be excluded if they meet any of the following criteria:

Have a known orthopedic or neurological condition.

Have a history of recent cervical or spinal surgery.

Have a diagnosed psychiatric disorder.

Have any medical contraindication to performing physical activity or exercise.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
The Extensor Endurance Test | baseline, immediately after the intervention
  The Extensor Endurance Test was conducted in prone position, with the participant asked to hold the head in a neutral position with the chin tucked. Time to fatigue (in seconds) was recorded for both tests
The Neck Flexor Endurance | baseline, immediately after the intervention
  The Neck Flexor Endurance Test was performed in a semi-supine position, with the participant instructed to lift and hold the head at 2.5 cm above the table surface until fatigue

SECONDARY OUTCOMES:
Neck Disability Index | baseline, immediately after the intervention
  The NDI consisted of 10 items assessing neck-related functional limitations, with a maximum score of 50, higher scores indicating greater disability.
Numeric Rating Scale | baseline, immediately after the intervention
  The NRS ranged from 0 (no pain) to 10 (worst imaginable pain) and was administered pre- and post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University, Karabük, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No